CLINICAL TRIAL: NCT00001155
Title: Treatment of Wegener's Granulomatosis With Cyclophosphamide
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 760042; 76-I-0042
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2002-02

CONDITIONS: Vasculitis; Wegener's Granulomatosis
Keywords: Vasculitis; Prednisone; Granuloma; Wegener's Granulomatosis; Cyclophosphamide; Renal Biopsy
MeSH Terms: conditions — Vasculitis; Granulomatosis with Polyangiitis; Granuloma | interventions — Cyclophosphamide

INTERVENTIONS:
Drug: cyclophosphamide

SUMMARY:
The purpose of this protocol is to continue to treat patients with Wegener's granulomatosis who have already entered the study, and to treat new patients. The investigators will attempt to correlate the clinical response with specific immunosuppressive effects of drug administration. The investigators are accumulating data on the optimal duration and side effects of therapy.

DETAILED DESCRIPTION:
The purpose of the protocol is to continue to treat patients with Wegener's granulomatosis who have already entered the study, and to treat new patients. The investigators will attempt to correlate the clinical response with specific immunosuppressive effects of drug administration. The investigators are accumulating data on the optimal duration and side effects of therapy.

Age Range: greater than 1 year

ELIGIBILITY:
Patients greater than 1 year of age with the clinical and pathological diagnosis of WG whose illness presents a risk of permanent disability or death. Examples of processes that impart risk of permanent disability or death include: peripheral and central nervous system disease, cardiac involvement, glomerulonephritis, and vascular comprise of gastrointestinal organs.

No women who are pregnant or intend to become pregnant.

No patients who have known malignancies.

Patients must be HIV negative.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200
Dates: Start 1976-02; Study Completion 2002-02

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Allergy and Infectious Diseases (NIAID), Bethesda, Maryland, United States

REFERENCES:
- [Background] Talar-Williams C, Hijazi YM, Walther MM, Linehan WM, Hallahan CW, Lubensky I, Kerr GS, Hoffman GS, Fauci AS, Sneller MC. Cyclophosphamide-induced cystitis and bladder cancer in patients with Wegener granulomatosis. Ann Intern Med. 1996 Mar 1;124(5):477-84. doi: 10.7326/0003-4819-124-5-199603010-00003. PMID 8602705
- [Background] Hoffman GS, Kerr GS, Leavitt RY, Hallahan CW, Lebovics RS, Travis WD, Rottem M, Fauci AS. Wegener granulomatosis: an analysis of 158 patients. Ann Intern Med. 1992 Mar 15;116(6):488-98. doi: 10.7326/0003-4819-116-6-488. PMID 1739240